CLINICAL TRIAL: NCT06637163
Title: A Randomized Controlled, Multicenter Clinical Study of Benmelstobart Combined With Radiochemotherapy Versus Radiochemotherapy as Neoadjuvant Treatment for Esophageal Squamous Cell Carcinoma
Brief Title: Benmelstobart Combined With Radiochemotherapy as Neoadjuvant Treatment Iin ESCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2024-236R
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-10

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Paclitaxel; Carboplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Benmelstobart combined with radiochemotherapy (Experimental): Benmelstobart + Paclitaxel + Carboplatin + Radiotherapy
  Interventions: Drug: Benmelstobart+ Paclitaxel + Carboplatin+ Radiotherapy
- radiochemotherapy (Active Comparator): Paclitaxel + Carboplatin + Radiotherapy
  Interventions: Drug: Paclitaxel + Carboplatin + Radiotherapy

INTERVENTIONS:
Drug: Benmelstobart+ Paclitaxel + Carboplatin+ Radiotherapy — Benmelstobart: 1200 mg, i.v.gtt , d1, 22; Paclitaxel 50mg/m2, i.v.gtt , d1, 8, 15, 22, 29; Carboplatin AUC 2 mg/mL per minute, i.v.gtt , d1, 8, 15, 22, 29; Radiotherapy 41.4 Gy in 23 fractions, 5 days per week(If the number of patients achieving pCR in this group is ≥ 18 with the first 30 patients enrolled, the subsequent 20 patients will receive a reduced dose of 36 Gy in 20 fractions, 5 days per week.)
  Arms: Benmelstobart combined with radiochemotherapy
Drug: Paclitaxel + Carboplatin + Radiotherapy — Paclitaxel 50mg/m2, i.v.gtt , d1, 8, 15, 22, 29; Carboplatin AUC 2 mg/mL per minute, i.v.gtt , d1, 8, 15, 22, 29; Radiotherapy 41.4 Gy in 23 fractions, 5 days per week
  Arms: radiochemotherapy

SUMMARY:
This study will explore the efficacy and safety of benmelstobart combined with radiochemotherapy compared to radiochemotherapy alone as neoadjuvant treatment for esophageal squamous cell carcinoma. It will also compare the effectiveness and safety of low-dose radiotherapy versus standard-dose radiotherapy in neoadjuvant regimens that include benmelstobart with concurrent radiochemotherapy. This research may provide more treatment options for patients with esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
Eligible participants will be randomly assigned in a 1:1 ratio to either the benmelstobart plus radiochemotherapy group or the radiochemotherapy group. Surgery will be performed 6-8 weeks after the completion of neoadjuvant treatment, with the primary endpoint being the rate of pathological complete response (pCR).

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily participate in this study and sign informed consent forms, with good compliance.
* Aged 18 years and older, regardless of gender.
* ECOG performance status: 0-1.
* Patients with histologically confirmed clinical stages T1-3N+M0 or T3NanyM0 of resectable esophageal squamous cell carcinoma.
* No prior antitumor treatment for esophageal cancer, including chemotherapy, hormone therapy, radiotherapy, or immunotherapy.
* Laboratory tests must meet the following criteria (within 7 days prior to baseline enrollment):

  1. Complete blood count: a. Hemoglobin (Hb) ≥ 90 g/L (no blood transfusion in the last 14 days); b. Neutrophil count (NEUT) ≥ 1.5 × 10^9/L; c. Platelet count (PLT) ≥ 100 × 10^9/L; d. White blood cell count (WBC) ≥ 3 × 10^9/L;
  2. Biochemical tests: a. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; b. Total bilirubin (TBIL) ≤ 1.5 × ULN; c. Serum creatinine (Cr) ≤ 1.5 × ULN (or creatinine clearance (CCr) ≥ 60 mL/min);
  3. Coagulation function: activated partial thromboplastin time (APTT), International normalized ratio (INR), prothrombin time (PT) ≤ 1.5 × ULN;
  4. Thyroid function: Thyroid-stimulating hormone (TSH) ≤ ULN (if abnormal, FT3 and FT4 levels should also be assessed; if FT3 and FT4 levels are normal, the patient can be enrolled);
  5. Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ 50%;
* Female participants must agree to use contraception (e.g., intrauterine device [IUD], contraceptive pills, or condoms) during the study and for 6 months after the study ends; a negative serum pregnancy test must be obtained within 7 days prior to enrollment, and participants must not be breastfeeding. Male participants must also agree to use contraception during the study and for 6 months after the study ends.

Exclusion Criteria:

Participants with any of the following criteria will be excluded from the study:

* Presence of other malignant tumors (except for previously cured basal cell carcinoma of the skin).
* Diagnosis of cervical esophageal cancer.
* Severe hypersensitivity reactions following the administration of other monoclonal antibodies.
* Any active autoimmune disease or history of autoimmune disease (such as, but not limited to: autoimmune hepatitis, interstitial pneumonia, enteritis, vasculitis, nephritis; asthma requiring bronchodilator intervention). However, patients with the following conditions may be included: vitiligo, psoriasis, alopecia that do not require systemic treatment, well-controlled type 1 diabetes, and hypothyroidism with normal thyroid function under replacement therapy.
* Use of immunosuppressants, systemic, or absorbable local hormone therapy to achieve immunosuppressive effects (doses > 10 mg/day of prednisone or equivalent), and continuing use within 2 weeks of the first dose.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
* Uncontrollable neurological symptoms from brain metastases, spinal cord compression, or carcinomatous meningitis occurring within 4 weeks prior to the first dose, or evidence of brain or leptomeningeal disease found on CT or MRI screening.
* Presence of any severe and/or uncontrolled disease, including:

  1. Acute or persistent myocardial ischemia or myocardial infarction, poorly controlled clinically significant arrhythmias, and NYHA class II or higher heart failure; LVEF < 50%.
  2. Active or uncontrolled severe infections (≥ CTCAE grade 2 infections).
* Vaccination with preventive or attenuated vaccines within 4 weeks prior to the first dose.
* Any factors, as judged by the investigator, that could lead to premature termination of the study, such as other serious illnesses (including mental illness) requiring concurrent treatment, significant laboratory abnormalities, or family or social factors that could affect participant safety.
* For participants who are HBsAg (+) and/or HBcAb (+), HBV DNA must be < 500 IU/mL (if the local center's lower limit of detection is higher than 500 IU/mL, the investigator may decide on enrollment based on specific circumstances) and must continue to receive effective anti-HBV treatment during the study, or must have initiated treatment with entecavir or tenofovir prior to the study drug.
* For participants who are HCV antibody positive, HCV-RNA testing is required; those with HCV-RNA > 10^3 copies/mL will be excluded.
* Positive HIV test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) | 4 months
  The ratio of patients with no residual cancer cells found in the pathological examination after treatment.

SECONDARY OUTCOMES:
Major pathologic response (MPR) | 4 months
  The percentage of subjects with a residual surviving tumor less than or equal to 10% after surgery.
Overall response rate (ORR) | 4 months
  The proportion of patients achieved a best overall tumor response of complete response (CR) or partial response (PR).
Diseases control rate (DCR) | 4 months
  The proportion of patients achieved CR+PR+ stable disease (SD).
R0 resection rate | 4 months
  The proportion of subjects who could undergo R0 resection.
Disease free survival (DFS), 1y-DFS | 15 months
  The time from surgery to the onset of tumor recurrence or death from any cause.
Overall survival (OS), 1y-OS | 15 months
  The time from randomization to the time of death from any cause.
Surgical-related Indicators | 1 months
  Surgical Time: Defined as the duration from the start to the end of the surgery for the participant.
  Intraoperative Blood Loss: Defined as the amount of blood lost by the participant during the surgery.
  Postoperative Length of Stay: Defined as the duration from the end of surgery until the participant is discharged.
  Perioperative Complication Rate: Defined as the percentage of participants who experience complications during the perioperative period among all participants.
Neoadjuvant Treatment Completion Rate | 1 months
  The percentage of participants who complete neoadjuvant treatment among all participants.
Adverse events | 15 months
  The severity of adverse events will be evaluated according to the NCI CTCAE 5.0 standard.

CONTACTS AND LOCATIONS:
Overall Officials: Lijie Tan, Professor, Principal Investigator — Fudan University
Locations (5):
- China (5):
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No